CLINICAL TRIAL: NCT02318082
Title: A Phase I Study of Individual Adult and Pediatric Patient Dose-escalated Interleukin-2 Therapy for Refractory Chronic Graft-versus-Host-Disease
Brief Title: Study of Individual Adult and Pediatric Patient Dose-escalated Interleukin-2 Therapy for Refractory Chronic GVHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-452
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Chronic Versus Graft Host Disease
Keywords: Chronic versus Graft Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interleukin-2 (IL-2) (Experimental): Interleukin-2: Each participant will receive daily subcutaneous IL-2 for self-administration per cycle. Each participant will start at Dose Level A. In the abscence of DLTs or severe non-DLT adverse events, participants will have daily SC IL-2 dose-escalated at Week 2 (to dose level B) and at Week 4 (to Dose Level C), and continue on their maximum tolerated dose (MTD) IL-2 for 4 weeks total.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2
  Other Names: Proleukin; Aldesleukin; IL-2

SUMMARY:
This research study is a way of gaining new knowledge about the treatment for cGVHD that has not responded to steroids. This research study is evaluating a drug called Interleukin-2 (IL-2) as a possible treatment for cGVHD. In this Phase I study, the investigators are looking to see if 8- week individual patient dose- escalated IL-2 therapy for cGVHD is safe and its effects on your immune cells.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved IL-2 for the treatment of cGVHD but it has been approved for metastatic renal cell carcinoma (MCC), and metastatic melanoma.

Chronic GVHD is a medical condition that may occur after the participant has received bone marrow, stem cell or cord blood transplant. The donor's immune system may recognize the participant's body (the host) as foreign and attempt to 'reject' it. This process is known as graft-versus-host-disease. Traditional standard therapy to treat cGVHD is prednisone (steroids). Interleukin-2 (IL-2) is a natural protein involved with regulation of white blood cells (WBCs). WBCs are part of the immune system.The investigators looking to see whether IL-2 helps control chronic GVHD by stopping the donor's immune system from 'rejecting' the participant's body.

This study will look to see if increasing the dose level of study drug every two weeks can be administered safely without severe or unmanageable side effects in participants that have cGVHD. Depending on how well you tolerate your initial dose level and subsequent dose levels, your study drug dose level may be increased a maximum of two times. These increases in dose levels will occur two weeks apart. All participants on the study will start at the same dose level.

Study Drug: You will administer, or have someone else administer if you are unable to yourself, IL-2 through an injection under your skin. You should rotate the injection site, if possible. You will do this once every day for 8- weeks.

During the first 8 weeks of IL-2, you will continue to take steroids and other immune suppressing medications without changing the dose your doctor has set for you while you are on IL-2. After 8 weeks of I L-2 therapy, your doctor may reduce the amount of steroids you take.

If your cGVHD improves after 8 weeks on dose-escalated IL-2, you may have the option of continuing extended duration therapy. Extended duration therapy is daily IL-2 treatment starting at the end of week 8. You will be re-assessed every 6 months while on extended duration IL-2 to determine if IL-2 therapy should continue, at the discretion of the treating physician.

Drug Diary: Each day of the first 8 weeks you take IL-2 and each day during extended-duration IL-2 (if applicable); you will be asked to document in a drug diary when you took the drug and where you injected it. The diary will also ask if the entire syringe was injected, and if there were other issues related to IL-2. You will be asked to return your drug diary to clinic every 2 weeks for the first 8 weeks of IL-2 and at least every 8 weeks for extended duration IL-2.

Chronic GVHD Assessments: While you are on study, a member of the study team will examine you to evaluate your cGVHD. These assessments may include examination of your skin, joints/muscles, eyes, mouth, lungs, and gastrointestinal system (for example, whether you have experienced any nausea, vomiting, diarrhea, difficulty swallowing). The investigators will also look at the range of motion of different body parts (for example, your arms).

ELIGIBILITY:
Inclusion Criteria

* Recipient of 7-8/8 HLA-matched (HLA-A, -B, -C, -DRB1) allogeneic hematopoietic stem cell transplantation
* Participants must have steroid-refractory cGVHD despite use of 2 or more agents. Steroid-refractory cGVHD is defined as having persistent signs and symptoms of cGVHD (Appendix C, D) despite the use of prednisone at ≥ 0.25 mg/kg/day (or 0.5 mg/kg every other day) for at least 4 weeks (or equivalent dosing of alternate glucocorticoids) without complete resolution of signs and symptoms. Participants with either extensive or limited chronic GVHD requiring systemic therapy are eligible.
* Stable dose of glucocorticoids for 4 weeks prior to enrollment.
* No addition or subtraction of other immunosuppressive medications (e.g., calcineurin-inhibitors, sirolimus, mycophenolate-mofetil) for 4 weeks prior to enrollment. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range of that drug.
* Participants must have adequate organ function as defined below:

  * Hepatic: Adequate hepatic function (total bilirubin ≤ 2.0 mg/dl-exception permitted in participants with Gilbert's Syndrome; AST (SGOT)/ALT (SGPT) ≤ 2x institutional ULN), unless hepatic dysfunction is a manifestation of presumed cGVHD. For participants with abnormal LFTs as the sole manifestation of cGVHD, documented GVHD on liver biopsy will be required prior to enrollment. Abnormal LFTs in the context of active cGVHD involving other organ systems may also be permitted if the treating physician documents the abnormal LFTs as being consistent with hepatic cGVHD, and a liver biopsy will not be mandated in this situation.
  * Pulmonary: FEV1 ≥ 50% or DLCO(Hb) ≥ 40% of predicted, unless pulmonary dysfunction is deemed to be due to chronic GVHD.
  * Renal: Serum creatinine ≤ institutional ULN or creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
  * Pediatric patients must have creatinine clearance ≥ 60 mL/min/1.73 m2 regardless of serum creatinine level.
  * Adequate bone marrow function indicated by absolute neutrophil count (ANC) ≥1000/mcL and platelets ≥ 50,000/mcL without growth factors or transfusions
  * Cardiac: No myocardial infarction within 6 months prior to enrollment or NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* Karnofsky/Lansky performance status ≥ 60% (Appendix A)
* Age ≥ 2 years. In our institutional experience and according to published reports, the incidence of cGVHD in children aged less than 2 years is rare. 41 Daily SC injections of low-dose IL-2 have been used in pediatric post-HSCT patients as young as 2 years. 39 Prolonged daily SC injections of other drugs such as low molecular weight heparin and insulin are commonly administered and well tolerated in the young pediatric population with the use of the Insuflon® indwelling SC catheter. The use of the Insuflon® indwelling SC catheter for IL-2 administration is not required for all pediatric patients and their use will depend on the preference of the patient and provider
* The effects of IL-2 on the developing human fetus are unknown. For this reason and because chemotherapeutic agents are known to be teratogenic, participants of child-bearing and child-fathering potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a female become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Males treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of IL-2 administration.
* Ability to understand and/or the willingness of participant or their parent/legally authorized representative to sign a written informed consent document.

Exclusion Criteria:

* Participants with ongoing prednisone (equivalent) dose requirement > 1 mg/kg/day (or equivalent).
* Participants with concurrent use of calcineurin-inhibitor plus sirolimus (either agent alone is acceptable).
* Participants with new immunosuppressive medication, extra-corporeal photopheresis or rituximab therapy initiated in the 4 weeks prior.
* Participant with post-transplant exposure to donor lymphocyte infusion (DLI), or T-cell or IL-2 targeted medication (e.g. ATG, alemtuzumab, basiliximab, denileukin diftitox) within 100 days prior.
* Other investigational drugs within 4 weeks prior to enrollment, unless cleared by the Principal Investigator. Previous fixed-dose IL-2 therapy that was discontinued prior to 4 weeks is permitted.
* Participants with active malignant relapse or recrudescence of their prior hematologic disorder.
* Participants with inability to comply with IL-2 treatment regimen.
* Organ transplant (allograft) recipient.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the agents used after allogeneic HSCT. In addition, these individuals are at increased risk of lethal infections. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to IL-2.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Individuals with active uncontrolled hepatitis B or C are ineligible as they are at high risk of lethal treatment-related hepatotoxicity after HSCT.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of 8-week Individual patient dose-escalated Interleukin-2 | 8 weeks
  Participants will be evaluated over the course of the 8-week treatment for Dose-Limiting Toxicities (DLTs) from the individual dose-escalated IL-2

SECONDARY OUTCOMES:
Overall cGVHD Clinical Response Rate | Baseline, 8 Weeks
  Participants will have their cGVHD evaulated at baseline and at 8 weeks using the NIH Consensus criteria
Overall Survival Rate | 1 year
  Participants will have overall survival assessed by 1 year after study entry and immunologic assessment during the 8-week treatment
Malignant Relapse Rate | 1 Year
  Participants will have malignant relapse rate assessed by 1 year after study entry and immunologic assessment during the 8-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, DPhil, MBBS, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Insitute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Whangbo JS, Kim HT, Mirkovic N, Leonard L, Poryanda S, Silverstein S, Kim S, Reynolds CG, Rai SC, Verrill K, Lee MA, Margossian S, Duncan C, Lehmann L, Huang J, Nikiforow S, Alyea EP 3rd, Armand P, Cutler CS, Ho VT, Blazar BR, Antin JH, Soiffer RJ, Ritz J, Koreth J. Dose-escalated interleukin-2 therapy for refractory chronic graft-versus-host disease in adults and children. Blood Adv. 2019 Sep 10;3(17):2550-2561. doi: 10.1182/bloodadvances.2019000631. PMID 31471324